CLINICAL TRIAL: NCT02876679
Title: Cyclophosphamide Versus Anti-thymocyte Globulin for GVHD Prophylaxis After RIC Allo-SCT
Acronym: ATG-CyGVHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P150955; 2016-002129-12 (EudraCT Number)
Record Dates: First submitted 2016-08-12; First posted 2016-08-24 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Graft vs Host Disease
Keywords: Hematopoietic Stem Cell; Transplantation; Graft vs Host Disease; Cyclophosphamide; Anti-Thymocyte Globulin; GVHD prophylaxis
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cyclophosphamide; Antilymphocyte Serum; Transplantation Conditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclophosphamide (Experimental): 50mg/Kg/day cyclophosphamide (day +3 and +4)
  Interventions: Drug: Cyclophosphamide; Drug: Conditioning regimen
- Anti-Thymocyte Globulin (Active Comparator): 2.5 mg/Kg/day ATG (Thymoglobuline®) for 2 consecutive days (day -2 and -1)
  Interventions: Drug: Anti-Thymocyte Globulin; Drug: Conditioning regimen

INTERVENTIONS:
Drug: Cyclophosphamide — GVHD prophylaxis: All patients will receive post-transplant 50mg/Kg/day cyclophosphamide (day +3 and +4) AND cyclosporine-A alone in case of an HLA-sibling donor, or cyclosporine-A and mycophenolate-mofetil in case of an HLA-matched unrelated donor
  Other Names: Cyclophosphamide + cyclosporine-A +/-mycophenolate-mofetil
  Arms: Cyclophosphamide
Drug: Anti-Thymocyte Globulin — GVHD prophylaxis: 2.5 mg/Kg/day ATG (Thymoglobuline®) for 2 consecutive days (day -2 and -1) All patients will receive cyclosporine-A alone in case of an HLA-sibling donor, or cyclosporine-A and mycophenolate-mofetil (MMF) in case of an HLA-matched unrelated donor.
  Other Names: Anti-Thymocyte Globulin + cyclosporine-A +/-mycophenolate-mofetil
  Arms: Anti-Thymocyte Globulin
Drug: Conditioning regimen — 30 mg/m2/day fludarabine for 5 days (day-6 to day-2) 130 mg/m2/day IV busulfan once daily for 2 days (day -4 and -3)

SUMMARY:
The study is designed as a two arm randomized Phase II, multicenter trial comparing cyclophosphamide to anti-thymocyte globulin for Graft-versus-Host Disease (GVHD) prophylaxis in patients with hematologic malignancies undergoing reduced intensity conditioning hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Allogeneic stem cell transplantation (allo-SCT) is a well-established therapy for different hematologic malignancies. Reduced-intensity conditioning (RIC) regimens can decrease the rate of toxicity/mortality in elderly patients, or in patients with poor medical condition. GVHD prophylaxis remains a challenging task after allo-SCT. The Flu-ivBu combination is a widely used RIC regimen, endorsed by EMA since July 2014. ATG in combination with cyclosporine-A ±mycophenolate mofetil is the backbone for GVHD prophylaxis in this setting. ATG can prevent GVHD with a good efficacy, but at the cost of a higher toxicity and profound immunosuppression, calling for more effective therapies. The most widely used RIC regimen in France incorporates fludarabine (Flu), intermediate doses of IV-busulfan (Bu) and anti-thymocyte globulins (ATG). While the use of ATG can prevent severe acute and chronic GVHD after allogeneic peripheral blood stem cell (PBSC) transplantation from both HLA-identical sibling and unrelated donors, some data suggested that in-vivo T-cell depletion with ATG in the RIC setting may induce a higher risk of disease relapse. Also, ATG induces profound immune suppression and increase incidence of opportunistic infections, especially EBV-related complications (relative risk=4.9; 95% CI[ 1.1-21.0]; P=0.03).

On the other hand, high-dose post-transplantation cyclophosphamide (PTCy) was developed to facilitate HLA-haploidentical allo-SCT using unmanipulated bone marrow (BM) cells. PTCy was effective in preventing both acute and chronic GVHD given its capacity to preferentially eliminate allo-reactive T cells and preserve regulatory T cells, both of which impact allogeneic immune reactions. Subsequently, the efficacy of PTCy as sole GVHD prophylaxis after myeloablative conditioning when using BM was also shown. However, BM is not the preferred source of stem cells after RIC allo-SCT, and the potential efficacy of PTCy on preventing GVHD when using PBSCs (which is the most frequently used source of allogeneic cells worldwide) is debated.

The advent of PTCy therapy is nowadays on the cutting edge. Thus, the potential efficacy (and cost-effectiveness) of PTCy for GVHD prophylaxis may have a major ATG sparing potential. A recent single centre phase 2 study (n=49) suggested that PTCy alone may not be the preferred GVHD prophylaxis following a RIC transplant with PBSCs. Indeed, A matched cohort analysis compared outcomes to tacrolimus/methotrexate GVHD prophylaxis and indicated higher rates of acute GVHD grade II to IV (46% versus 19%; hazard ratio [HR], 2.8; P =0.02) and treatment-related mortality (HR, 3.3; P =0.035) and worse overall survival (HR, 1.9; P=0..04) with post-CY. Interpretation of the above non-randomized data is further complicated by heterogeneity (related and unrelated donors, BM and PBSC as stem cell source, different conditioning regimen), highlighting the need for a controlled randomized trial in a standardized setting.

The ultimate goal of this Phase IIB study is to assess the feasibility and inform the design of a subsequent phase III study. The present randomized trial is designed to compare the efficacy of the addition of PTCy to current standard of care with ATG after a Flu-Bu-based RIC regimen on GVHD prophylaxis. The protocol will use a novel endpoint for benchmarking interventions based on a composite primary endpoint of GVHD-free, relapse-free survival which measures freedom from ongoing morbidity and represents an ideal outcome measure after allo-SCT.

ELIGIBILITY:
Inclusion Criteria :

* Patients aged between 18 and 65 years
* Presence of a hematologic malignancy for which a reduced-intensity conditioning allo-SCT is indicated (eligibility criteria for RIC allo-SCT include at least one of the following parameters: (i) patient age older than 50 years; (ii) heavily pre-treated patients who received an autologous hematopoietic SCT (auto-SCT) or with more than 2 lines of chemotherapy before allo-SCT; and (iii) patients with poor performance status because of significant medical comorbidities as described by Sorror et al.
* Karnofsky index ≥ 70%
* Availability of a sibling or unrelated stem-cell donor (10/10-HLA matched unrelated donor)
* Efficient contraceptive method within 1 month for women and 3 months for men after the last dose of treatment
* Written informed consent.

Exclusion Criteria:

* Creatinine clearance less than 30 mL/min
* Bilirubin or amino-transferases above 3X upper normal limit
* Cardiac ejection fraction less than 40%
* Pulmonary impairment with <50% lung carbon monoxide diffusing capacity (DLCO)
* Known hypersensitivity or contraindication to the use of post-transplant Cy and ATG
* Any circumstance that precludes the use of the drugs involved in the protocol
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of GVHD-free, relapse-free survival (GRFS) | 12 Months
  Absence of grade 3-4 acute GVHD, chronic GVHD requiring systemic treatment, relapse, or death

SECONDARY OUTCOMES:
Cumulative incidence of grade 2-4 and grade 3-4 severe acute GVHD | 6 Months
  Acute GVHD grading should be performed by the revised Glucksberg criteria (Przepiorka et al., 1995). The time of onset of acute grades II-IV and III-IV acute GVHD will be recorded, as well as the maximum grade achieved
Cumulative incidence of non-relapse mortality within the first 12 months after transplantation. | 12 Months
  Death without evidence of disease recurrence. Disease recurrence will be considered a competing event.
Disease-free survival | 12 months
  Relapse-free survival : time from date of transplant to death or relapse, whichever comes first. The event for this endpoint is relapse or death. Patients alive and free from disease relapse will be censored at last follow-up
Overall survival. | 12 months
  Overall survival : time interval between date of transplant and death from any cause or for surviving patients, to last follow-up. The event for this endpoint is death from any cause.
Quality of Life (QoL) with EORTC QLQ-C30 | 12 Months
  Evaluation by the questionnaire EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30)
Quality of Life (QoL) with FACT-BMT | 12 Months
  Evaluation by the questionnaire FACT-BMT (Functional Assessment of Cancer Therapy - Bone Marrow Transplant)
Immune recovery measurement | 12 Months
  Immune recovery measurement: number of patients with complete immune recovery (T, B and dendritic cells subsets)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad MOHTY, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Saint Antoine Hospital - Hematology Department, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brissot E, Labopin M, Labussiere H, Fossard G, Chevallier P, Guillaume T, Yakoub-Agha I, Srour M, Bulabois CE, Huynh A, Chantepie S, Menard AL, Rubio MT, Ceballos P, Dulery R, Furst S, Malard F, Blaise D, Mohty M. Post-transplant cyclophosphamide versus anti-thymocyte globulin after reduced intensity peripheral blood allogeneic cell transplantation in recipients of matched sibling or 10/10 HLA matched unrelated donors: final analysis of a randomized, open-label, multicenter, phase 2 trial. Blood Cancer J. 2024 Feb 19;14(1):31. doi: 10.1038/s41408-024-00990-3. PMID 38374026
- [Derived] Del Pozo Martin Y. 47th Annual Meeting of the EBMT. Lancet Haematol. 2021 May;8(5):e317-e318. doi: 10.1016/S2352-3026(21)00104-6. Epub 2021 Mar 31. No abstract available. PMID 33811823